CLINICAL TRIAL: NCT00744965
Title: A Randomized Controlled Clinical Trial of Treatment of Mild Gestational Diabetes With Glyburide Versus Placebo
Brief Title: Treatment of Mild Gestational Diabetes With Glyburide Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Leveno, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 032011-086; 042008-058 (Other: UTexasSouthwestern); NCT00942552 (obsolete NCT alias)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Mild Gestational Diabetes
MeSH Terms: interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glyburide (Active Comparator): Women with mild gestational diabetes will be started ADA diet and a low dose of Glyburide and their medication dosage will be titrated as necessary during the pregnancy to achieve glucose control.
  Interventions: Drug: Glyburide
- Placebo (Placebo Comparator): Women with mild gestational diabetes will be started ADA diet and placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glyburide — Starting dosage is 2.5 mg once daily. This dose will be titrated as necessary during the pregnancy to achieve glycemic control.
  Arms: Glyburide
Drug: Placebo — Sham dose adjustments of the placebo will be made.
  Arms: Placebo

SUMMARY:
This is a randomized prospective trial which addresses the question of whether use of an oral hypoglycemic agent as an adjunct to diet therapy in women with mild gestational diabetes will result in achieving euglycemia in a shorter period of time and, in turn, result in less frequent maternal and neonatal morbidities. This study is designed to test the hypothesis that in women with mild GDM, use of Glyburide in addition to diet and nutritional counseling lowers mean infant birth weight by 200 grams as compared with diet and nutritional counseling alone.

ELIGIBILITY:
Inclusion Criteria:

* A glucose value of ≥140 mg/dl on a 50-gram oral glucose loading test by plasma at gestational age between 24 weeks 0 days and 27 weeks 6 days based on clinical information
* An Abnormal 3-hour oral glucose tolerance test with a fasting glucose of ≤105 mg/dl
* Gestational age of less than or equal to 28 weeks and 0 days at the time of consent/randomization
* Singleton gestation

Exclusion Criteria:

* Established pregestational diabetes
* Abnormal gestational diabetes testing (≥140) prior to 24 weeks 0 days of gestation. Women who have a negative glucose loading test (<140mg/dl) before 24 weeks may still be considered for this study if they present again for glucose tolerance testing between 24 and 27 weeks.
* Multiple gestations
* Known major fetal anomaly or fetal demise
* Any renal disease with serum creatinine of >1.0
* Known liver disease such as hepatitis
* Maternal or fetal conditions likely to require imminent or very preterm delivery such as preeclampsia, preterm premature rupture of the membranes, preterm labor, and intrauterine fetal growth restriction
* Known hypersensitivity or allergic reaction to Glyburide

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 395 (Actual)
Dates: Start 2008-09-16 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Result] Casey BM, Duryea EL, Abbassi-Ghanavati M, Tudela CM, Shivvers SA, McIntire DD, Leveno KJ. Glyburide in Women With Mild Gestational Diabetes: A Randomized Controlled Trial. Obstet Gynecol. 2015 Aug;126(2):303-309. doi: 10.1097/AOG.0000000000000967. PMID 26241419

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Glyburide
Started | 197 | 198
Completed | 186 | 189
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glyburide | Placebo | Total
Number analyzed (Participants) | 189 | 186 | 375
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 189 | 186 | 375
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (6) | 31.2 (6) | 31.2 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 186 | 375
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 189 | 186 | 375

OUTCOME MEASURES:

1. Primary Outcome: Mean Fetal Weight at Birth
Time Frame: Immediately after delivery of fetus
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
grams | 3355 (521) | 3322 (481)

2. Secondary Outcome: Number of Participants With Large for Gestational Age Infants
Description: Birth weight exceeding the 90th percentile for the gestational age at delivery.
Time Frame: After delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 22 | 20

3. Secondary Outcome: Macrosomia
Description: birth weight 4,000 g or greater
Time Frame: After delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 18 | 13

4. Secondary Outcome: Neonatal Intensive Care Unit Admissions
Time Frame: Until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 11 | 13

5. Secondary Outcome: Rate of Cesarean Delivery
Time Frame: After delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 67 | 70

6. Secondary Outcome: Diagnosis of Pregnancy-induced Hypertension
Time Frame: until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 12 | 15

7. Secondary Outcome: Shoulder Dystocia
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 1 | 0

8. Secondary Outcome: Need for Insulin Treatment
Time Frame: after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 4 | 4

9. Secondary Outcome: 3rd or 4th Degree Perineal Laceration
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 5 | 1

10. Secondary Outcome: Chorioamnionitis
Description: Maternal fever >=38.0°C
Time Frame: intrapartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 12 | 15

11. Secondary Outcome: Need for Insulin Therapy
Time Frame: throughout pregnancy and delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Glyburide
Number analyzed (Participants) | 186 | 189
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: approximately 3-4 months (throughout the duration of study participation)
Arm/Group | Placebo | Glyburide
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/189
Serious Adverse Events (participants affected / at risk) | 0/186 | 1/189
Other Adverse Events (participants affected / at risk) | 0/186 | 0/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=186) | Glyburide (N=189)
facial swelling (Endocrine disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size of 395 limits our ability to analyze the effect of Glyburide on uncommon pregnancy outcomes. The study was underpowered for outcomes other than birth weight difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No